CLINICAL TRIAL: NCT01491308
Title: Restrictive Versus Liberal Red Cell Transfusion Strategy in Orthopedic-Oncology Patients Undergoing Surgery - a Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMAC-11-IM-0449-11-CTIL
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Red Blood Cells Transfusion.

ARMS (2):
- Restrictive (Active Comparator): Hemoglobin concentrations will be maintained in the range of 7.5 to 9.0 g per deciliter, with a transfusion given when the hemoglobin concentration is below 7.5 g per deciliter.
  Interventions: Other: Red blood cells transfusion
- Liberal (Active Comparator): Hemoglobin concentrations will be maintained in the range of 10.0 to 12.0 g per deciliter, with a transfusion given when the hemoglobin concentration is below 10.0 g per deciliter.
  Interventions: Other: Red blood cells transfusion

INTERVENTIONS:
Other: Red blood cells transfusion — This transfusion policy holds to any time from the start of surgery until discharge. The physicians caring for the patient will be instructed to administer transfusion, one unit at a time, and to measure the patient's hemoglobin concentration after each unit is transfused. In both groups, no further units will be given if the goal hemoglobin was obtained (7.5 g per deciliter for the restrictive arm and 10.0 g per deciliter for the liberal one). All other management decisions are left to the discretion of the patients' physicians. Attending physicians can administer RBC transfusions outside the rules of the protocol (i.e more than 1 unit at a time, without determining pre-transfusion hemoglobin) if severe acute bleeding occurs or other forms of circulatory shock.

SUMMARY:
The rationale for perioperative red blood cell (RBC) transfusion is based on the observation that anemia is an independent risk factor for morbidity and mortality after cardiac operations. However, transfusions have been associated with high rates of morbidity and mortality in critically ill patients, and some recent studies have shown worse outcomes, including increased occurrence of renal failure and infection, as well as respiratory, cardiac, and neurological complications, in transfused compared with non transfused patients after cardiac surgery. On the basis of past clinical observations, some authors have suggested that hematocrit should be maintained at around 30% and hemoglobin concentration at 10 g/dL. Recently, however, this hemoglobin threshold has been reconsidered because of recognized risks associated with transfusion and greater appreciation of the importance of individual physiological responses to anemia. In a comparative trial of 428 patients undergoing elective coronary artery bypass graft(CABG) surgery, Bracey et al reported that reducing the hemoglobin trigger to 8 g/dL did not adversely affect patient outcomes and resulted in lower costs. An important multicenter Canadian Study by Hebert et al that included a large number of critically ill patients revealed that A restrictive strategy of red-cell transfusion (hemoglobin concentration maintained between 7.0and 9.0g/dL) is at least as effective as and possibly superior to a liberal transfusion (hemoglobin concentration between 10 and 12 g/dL) strategy in critically ill patients, with the possible exception of patients with acute myocardial infarction and unstable angina, in terms of reducing organ dysfunction and mortality.

The investigators would like to determine whether a restrictive strategy of red-cell transfusion and a liberal strategy produce equivalent results in orthopedic-oncology patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive ASA I-III patients, with preoperative hemoglobin 12 gr% or less scheduled for major orthopedic-oncology surgery (one that is expected to carry moderate to severe blood loss) at Tel Aviv Sourasky Medical Center will be included in the study.

Exclusion Criteria:

* Patients will be excluded for any of the following reasons:
* an age of less than 18 years;
* inability to receive blood products;
* pregnancy;
* emergency procedures;
* hepatic dysfunction (total bilirubin value higher than 1.5 mg/d);
* end-stage renal disease (receiving chronic dialysis therapy);
* acute coronary syndrome, active heart or lung disease and refusal to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 6 weeks post surgery
  Functional outcome during hospital stay and at 6 weeks as defined by the Modified Rivermead Mobility Index attached below (a functional index that measures different functionalities of the patient. This index is daily measured by the physiotherapist's group
Mortality and morbidity | 6 weeks post surgery
  A composite end point that includes all cause mortality and morbidity occurring till 6 weeks post surgery.

SECONDARY OUTCOMES:
Admission to ICU | 6 weeks post surgery
Hospital lengths of stay | 6 weeks post surgery
RBC transfusions | Hospitaliztion
  The investigators will also evaluate the incidence of RBC transfusions and the number of units transfused.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066